CLINICAL TRIAL: NCT00673010
Title: Lesion Dosimetry With 124-Iodine in Metastatic Thyroid Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-116
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Thyroid Cancer
Keywords: 124-IODINE; I-131 METAIODOBENZ SULF (MIBG); Thyroid; Parathyroid
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases | interventions — Iodine-131

ARMS (1):
- 1 (Experimental): 131 I-iodine (131-I), 124 I-iodine (124-I)
  Interventions: Radiation: 131 I-iodine (131-I), 124 I-iodine (124-I)

INTERVENTIONS:
Radiation: 131 I-iodine (131-I), 124 I-iodine (124-I) — Those who have demonstrated metastases which concentrate radioiodine will undergo routine testing to determine the MTA for blood and lung tissue. This will be performed with 124-I instead of 131-I. If the diagnostic scans (done with 123-I) show that the metastatic lesions concentrate radioiodine, the patient will be treated with 131-I based on standard of care discussions at a tumor board meeting. One week following the 131-I therapy, a whole body scan will be obtained and compared with the 124-I diagnostic scan. One year later, another extent of disease workup will be performed which will include 124-I dosimetry and scanning.

SUMMARY:
One of the most effective treatments for metastases from thyroid cancer is a form of radioactive iodine known as 131-I. For more than 50 years, 131-I has been used to find and destroy thyroid cancer cells that have spread to other parts of the body. In many cases this treatment destroys the metastatic cells. However, in some patients it does not appear to work completely. This study is designed to use a slightly different form of radioactive iodine (called 124-I) which can precisely predict the amount of radiation that each metastatic lesion will receive.

124-I was developed at Memorial Sloan-Kettering in the 1950s and has been used here and at many other medical centers around the world for diagnostic studies. It has been found to be very safe and effective at finding metastatic lesions. The high resolution of newer PET scanners now allows us to carefully determine how much radiation each metastatic lesion will receive. If 124-I can accurately predict which patients will not respond to 131-I treatments we can then avoid exposing those patients to unnecessary radiation. For the rest of the patients we can custom tailor the 131-I dose to destroy the metastatic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Adult thyroid carcinoma patients who have had a total thyroidectomy, histology confirmed by an MSKCC attending pathologist, and radioiodine remnant ablation.
* Adult thyroid carcinoma patients who have previously demonstrated radioiodine-avid metastases and are about to undergo Thyrogen-assisted dosimetry at MSKCC.
* The patient and physician are planning to administer 131-I for therapy if persistent radioiodine-avid metastases are present.
* Men and women of all races, ethnicities, and religious backgrounds are eligible.
* All subjects must have measurable disease, documented within the previous six months by ultrasonography (US), MRI, or non-contrast CT scanning.

Exclusion Criteria:

* Thyroid cancer patients who do not have metastases.
* Thyroid cancer patients who have not demonstrated that their metastases concentrate radioiodine.
* Patients who are under therapy for other active cancers.
* Anaplastic or Medullary thyroid carcinoma.
* Age less than 18 years.
* Patient who have received a therapeutic dose of radioiodine within the preceding nine months will not be eligible.
* Patients who plan to withdraw from thyroid hormone prior to dosimetry.
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-03-07 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
To estimate the relationship between the radiation dose and response to radiation at one year for metastatic lesions arising from differentiated thyroid carcinoma, following a single therapeutic administration of 131-Iodine. | conclusion of the study

SECONDARY OUTCOMES:
To determine the diagnostic sensitivity of the 124-Iodine whole body scan based on the 131-Iodine post-therapy scan (the "gold-standard"). | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Grewal, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org